CLINICAL TRIAL: NCT06662201
Title: Association Between P0.1 and Extubation Failure in Adult Patients with Acute Hypoxemic Respiratory Failure. a Multicenter Prospective Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Argentinian Intensive Care Society (Other)
Responsible Party: Sponsor
Other Study IDs: P01
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-09

CONDITIONS: Ventilator Weaning
Keywords: Respiration, artificial; Positive-Pressure Respiration
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acute respiratory failure: Adult patients (over 17 years of age) who have been intubated for acute respiratory failure hypoxemia for more than 24 hours, who have overcome a spontaneous breathing trial (SBT) and are fit to be extubated in the intensive care unit of the participating centers, who meet the inclusion criteria, who do not have exclusion criteria and from whom informed consent is obtained (from them or their immediate family member).

SUMMARY:
The goal of this observational study is to learn about the effect of the occlusion pressure during the first 100 miliseconds (P01) over the extubation failure in participants receiving mechanical ventilation for acute respiratory failure.

The main question it aims to answer is:

Are high P0.1 values (≥3 cmH2O) measured 30 minutes after starting a spontaneous breathing trial associated with extubation failure in adult patients who were intubated for acute hypoxemic respiratory failure?

ELIGIBILITY:
Inclusion Criteria:

* Patients over 17 years of age
* Patients receiving invasive mechanical ventilation for more than 24 hours
* Patients who have been ventilated for acute hypoxemic respiratory failure
* Patients who overcome a PVE
* Patients who, after overcoming the PVE, meet the conditions to be extubated immediately after, according to the team of treating professionals who conduct the weaning
* Patients who are in their first attempt at extubation

Exclusion Criteria:

* Tracheostomized patients
* Patients with neuromuscular disease (For example: Guillain Barré,
* Myasthenia Gravis, Amyotrophic lateral sclerosis, etc.)
* Patients with a decision not to reintubate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (over 17 years of age) who have required intubation and connection to mechanical ventilation due to acute respiratory failure hypoxemia for more than 24 hours, who have overcome a PVE and are ready to be extubated in the Intensive Care Units of the metropolitan area of Buenos Aires (AMBA).
Sampling Method: Non-Probability Sample
Enrollment: 256 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-08-29 (Estimated)

PRIMARY OUTCOMES:
Extubation failure | From enrollment to the end of follow-up at day 7
  Extubation failure is defined as reintubation by day 7. The decision to reintubate a patient will be made by the treating team, who will be blinded to the P0.1 values measured during spontaneus breathing trial.

SECONDARY OUTCOMES:
Cut-off point of P01 | From enrollment to the end of follow-up at day 7
  To identify the best cut-off point of P0.1 to predict extubation failure in adult patients who required invasive mechanical ventilation for acute hypoxemic respiratory failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanatorio Anchorena Recoleta, Buenos Aires, Buenos Aires F.D., Argentina

REFERENCES:
- [Background] Fernandez R, Raurich JM, Mut T, Blanco J, Santos A, Villagra A. Extubation failure: diagnostic value of occlusion pressure (P0.1) and P0.1-derived parameters. Intensive Care Med. 2004 Feb;30(2):234-240. doi: 10.1007/s00134-003-2070-y. Epub 2003 Nov 8. PMID 14608459
- [Background] Thille AW, Gacouin A, Coudroy R, Ehrmann S, Quenot JP, Nay MA, Guitton C, Contou D, Labro G, Reignier J, Pradel G, Beduneau G, Dangers L, Saccheri C, Prat G, Lacave G, Sedillot N, Terzi N, La Combe B, Mira JP, Romen A, Azais MA, Rouze A, Devaquet J, Delbove A, Dres M, Bourenne J, Lautrette A, de Keizer J, Ragot S, Frat JP; REVA Research Network. Spontaneous-Breathing Trials with Pressure-Support Ventilation or a T-Piece. N Engl J Med. 2022 Nov 17;387(20):1843-1854. doi: 10.1056/NEJMoa2209041. Epub 2022 Oct 26. PMID 36286317
- [Background] Sato R, Hasegawa D, Hamahata NT, Narala S, Nishida K, Takahashi K, Sempokuya T, Daoud EG. The predictive value of airway occlusion pressure at 100 msec (P0.1) on successful weaning from mechanical ventilation: A systematic review and meta-analysis. J Crit Care. 2021 Jun;63:124-132. doi: 10.1016/j.jcrc.2020.09.030. Epub 2020 Sep 30. PMID 33012587
- [Background] Spinelli E, Mauri T, Beitler JR, Pesenti A, Brodie D. Respiratory drive in the acute respiratory distress syndrome: pathophysiology, monitoring, and therapeutic interventions. Intensive Care Med. 2020 Apr;46(4):606-618. doi: 10.1007/s00134-020-05942-6. Epub 2020 Feb 3. PMID 32016537
- [Background] Alberti A, Gallo F, Fongaro A, Valenti S, Rossi A. P0.1 is a useful parameter in setting the level of pressure support ventilation. Intensive Care Med. 1995 Jul;21(7):547-53. doi: 10.1007/BF01700158. PMID 7593895
- [Background] Telias I, Damiani F, Brochard L. The airway occlusion pressure (P0.1) to monitor respiratory drive during mechanical ventilation: increasing awareness of a not-so-new problem. Intensive Care Med. 2018 Sep;44(9):1532-1535. doi: 10.1007/s00134-018-5045-8. Epub 2018 Jan 19. No abstract available. PMID 29350241
- [Background] Whitelaw WA, Derenne JP, Milic-Emili J. Occlusion pressure as a measure of respiratory center output in conscious man. Respir Physiol. 1975 Mar;23(2):181-99. doi: 10.1016/0034-5687(75)90059-6. PMID 1144940
- [Background] MacIntyre NR, Cook DJ, Ely EW Jr, Epstein SK, Fink JB, Heffner JE, Hess D, Hubmayer RD, Scheinhorn DJ; American College of Chest Physicians; American Association for Respiratory Care; American College of Critical Care Medicine. Evidence-based guidelines for weaning and discontinuing ventilatory support: a collective task force facilitated by the American College of Chest Physicians; the American Association for Respiratory Care; and the American College of Critical Care Medicine. Chest. 2001 Dec;120(6 Suppl):375S-95S. doi: 10.1378/chest.120.6_suppl.375s. No abstract available. PMID 11742959
- [Background] Ely EW, Baker AM, Dunagan DP, Burke HL, Smith AC, Kelly PT, Johnson MM, Browder RW, Bowton DL, Haponik EF. Effect on the duration of mechanical ventilation of identifying patients capable of breathing spontaneously. N Engl J Med. 1996 Dec 19;335(25):1864-9. doi: 10.1056/NEJM199612193352502. PMID 8948561
- [Background] Thille AW, Harrois A, Schortgen F, Brun-Buisson C, Brochard L. Outcomes of extubation failure in medical intensive care unit patients. Crit Care Med. 2011 Dec;39(12):2612-8. doi: 10.1097/CCM.0b013e3182282a5a. PMID 21765357
- [Background] Yu H, Luo J, Ni Y, Hu Y, Liu D, Wang M, Liang B, Liang Z. Early prediction of extubation failure in patients with severe pneumonia: a retrospective cohort study. Biosci Rep. 2020 Feb 28;40(2):BSR20192435. doi: 10.1042/BSR20192435. PMID 31990295
- [Background] Ionescu F, Zimmer MS, Petrescu I, Castillo E, Bozyk P, Abbas A, Abplanalp L, Dogra S, Nair GB. Extubation Failure in Critically Ill COVID-19 Patients: Risk Factors and Impact on In-Hospital Mortality. J Intensive Care Med. 2021 Sep;36(9):1018-1024. doi: 10.1177/08850666211020281. Epub 2021 Jun 2. PMID 34074160
- [Background] Dorado JH, Navarro E, Plotnikow GA, Gogniat E, Accoce M; EpVAr Study Group. Epidemiology of Weaning From Invasive Mechanical Ventilation in Subjects With COVID-19. Respir Care. 2023 Jan;68(1):101-109. doi: 10.4187/respcare.09925. Epub 2022 Nov 15. PMID 36379638
- [Background] Thille AW, Cortes-Puch I, Esteban A. Weaning from the ventilator and extubation in ICU. Curr Opin Crit Care. 2013 Feb;19(1):57-64. doi: 10.1097/MCC.0b013e32835c5095. PMID 23235542
- [Background] Pham T, Heunks L, Bellani G, Madotto F, Aragao I, Beduneau G, Goligher EC, Grasselli G, Laake JH, Mancebo J, Penuelas O, Piquilloud L, Pesenti A, Wunsch H, van Haren F, Brochard L, Laffey JG; WEAN SAFE Investigators. Weaning from mechanical ventilation in intensive care units across 50 countries (WEAN SAFE): a multicentre, prospective, observational cohort study. Lancet Respir Med. 2023 May;11(5):465-476. doi: 10.1016/S2213-2600(22)00449-0. Epub 2023 Jan 21. PMID 36693401